CLINICAL TRIAL: NCT03639337
Title: Use of Probiotics Bifidobacterium Longum, Bifidobacterium Breve and Bifidobacterium Infantis in Treating Pediatric Food Allergy to Milk or Egg.
Brief Title: Colonization and Persistence Capacity of a Multi-strain Probiotics in Pediatric Food Allergy to Milk or Egg.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Alessandro Giovanni Fiocchi, Director Clinical Research, Bambino Gesù Hospital and Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 787_OPBG_2014
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Food Hypersensitivity; Probiotic
Keywords: Probiotic; Food allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Allergic Children (Experimental): Allergic children to milk or egg, aged between 10 and 14 months, confirmed by double-blind oral provocation test against placebo.
  Intervention: 30 days of administration of multi-strain probiotics containing 3.5 x 109 UFC of Bifidobacterium longum BB536, Bifidobacterium breve M-16V and Bifidobacterium infantis M-63
  Interventions: Dietary Supplement: Multi-strain probiotic
- Not confirmed Allergic Children (No Intervention): Sensible children to milk or egg, aged between 10 and 14 months, not confirmed by double-blind oral provocation test against placebo.
- Controls (No Intervention): Healthy controls ages between 10 and 14 months

INTERVENTIONS:
Dietary Supplement: Multi-strain probiotic — 30 days of administration of multi-strain probiotics containing 3.5 x 109 UFC of Bifidobacterium longum BB536, Bifidobacterium breve M-16V and Bifidobacterium infantis M-63
  Arms: Allergic Children

SUMMARY:
This study evaluates the addition of three probiotics (Bifidobacterium longum, Bifidobacterium breve and Bifidobacterium infantis) in the treatment of pediatric food allergic children to milk or egg. The allergic participants will receive the probiotics, while other two populations age and sex matched of not confirmed allergic and healthy children will not receive probiotics.

DETAILED DESCRIPTION:
This study evaluates the colonization capacity of three probiotics (Bifidobacterium longum, Bifidobacterium breve and Bifidobacterium infantis) in milk and/or egg allergic children.

It is expected the recruitment of about 20 egg and/or milk allergic patients aged between 10 and 14 months old confirmed with double-blind oral tolerance test against placebo (Group 1).

Furthermore, about 10 patients sensible to milk or egg but not confirmed with double-blind oral tolerance test against placebo (Group 2) will be recruited and about 10 healthy individuals (Group 3).

For all 40 patients:

1. Baseline presence of Bifidobacterium longum BB536, Bifidobacterium breve M-16V and Bifidobacterium infantis M-63 will be evaluated;

   Only for Group 1 children it will be also evaluate:
2. The presence of the same strains during 30 days of administration of multi-strain probiotics containing 3.5 x 109 UFC of Bifidobacterium longum BB536, Bifidobacterium breve M-16V and Bifidobacterium infantis M-63 and after 60 days from the suspension of the administration.

Quantification of B. breve, B. longum subsp. longum and B. longum subsp. infantis in faecal samples was carried out by qRT-PCR using the Light Cycler 480 platform (Roche Diagnostics, Mannheim, Germany). The assays were performed with a 20 µl PCR amplification mixture containing: 10 µl LightCycler 480 Probe Master mix (Roche Diagnostics), 2 µl primers and probes (optimized concentrations, 0.5 µM and 0.1 µM, respectively), 3 µl molecular-grade H2O and 5 µl DNA template. Each sample was tested in duplicate to ensure data reproducibility. The RT-PCR temperature profile consisted of an initial denaturation at 95°C for 10 min, 45 amplification cycles at 95°C for 10 sec, 60°C for 30 sec and 72°C for 1 sec followed by a final cooling step at 40°C for 30 sec. Absolute quantification was performed using the "second derivative maximum method"

Statistical analyses: Wilcoxon signed-rank test was used to compare probiotic species concentrations during the time-course.

ELIGIBILITY:
Inclusion Criteria:

- Age between 10 and 14 months

Exclusion Criteria:

* gastrointestinal disease in progress or appearance in the last 30 days
* metabolic diseases
* antibiotic treatment in the 2 weeks prior to the start of the study;
* intake of probiotic, fermented milk or other functional foods in the two weeks preceding the start of the study.

Ages: 10 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2015-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Basal stool concentration of Bifidobacterium longum BB536, Bifidobacterium breve M-16V | 2 years
  It will be indicated number of cells per ul of stool.

SECONDARY OUTCOMES:
Stool concentration of Bifidobacterium longum BB536, Bifidobacterium breve M-16V after multi-strain probiotic administration. | 2 years
  It will be indicated number of cells per ul of stool.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Fiocchi, M.D., Principal Investigator — agiovanni.fiocchi@opbg.net
Locations (1):
- Ospedale Pediatrico Bambino Gesù, Roma, Italy